CLINICAL TRIAL: NCT04976764
Title: Affiliated Hospital of Qingdao University
Brief Title: The Correlation Between Cirrhotic Cardiomyopathy and Perioperative Cardiovascular Events in Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Other Study IDs: QYFYWZLL26462
Record Dates: First submitted 2021-07-15; First posted 2021-07-26 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Cirrhosis, Liver
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- liver cirrhosis with cirrhotic cardiomyopathy
- liver cirrhosis without cirrhotic cardiomyopathy

INTERVENTIONS:
Other:

SUMMARY:
Liver transplantation is an effective treatment for end-stage liver disease. Cardiovascular complications are the common causes of death in liver transplant recipients. The presence of cirrhosis cardiomyopathy has a potential impact on the prognosis of liver transplant recipients. Therefore, it is important to identify the high risk factors with cirrhotic cardiomyopathy before transplantation, so as to intervene earlier and improve the prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnostic criteria for decompensated liver cirrhosis: according to the guidelines for diagnosis and treatment of liver cirrhosis in 2019;
2. Diagnostic criteria for cirrhotic cardiomyopathy: in accordance with the revised criteria of CCM of international multidisciplinary Alliance for cirrhotic cardiomyopathy in 2019, the preoperative echocardiographic images of all patients were reviewed, and the systolic and diastolic dysfunction of all patients were evaluated.

Exclusion Criteria:

1. the compensatory liver cirrhosis, primary liver cancer without liver cirrhosis
2. Multiple organ transplantation or multiple organ transplantation
3. The preoperative echocardiographic data were not fully recorded, so that the exact diagnosis could not be made
4. There was no follow-up data or baseline data

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, the patients with decompensated liver cirrhosis who received liver transplantation from January 1, 2012 to June 1, 2021 in the Affiliated Hospital of Qingdao University were reviewed through the Yidu cloud platform. According to the 2019 cirrhosis cardiomyopathy (CCM) diagnostic criteria, they were divided into two groups according to the presence or absence of cardiomyopathy.The incidence of CCM , the predictive factors of perioperative and postoperative cardiovascular complications were followed up. At the same time,we analysed the influence of CCM on the survival rate.
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
perioperative cardiovascular events | 2012.1.1-2022.8
  there are differences between 2 groups.

IPD SHARING:
Plan to Share IPD: No